CLINICAL TRIAL: NCT03430908
Title: Blind Gastric Tube Placement: Incidence of Malposition Confirmed by Ultrasonography
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-653
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Anesthesia
Keywords: endotracheal tube; gastric tube; 17-653; Memorial Sloan Kettering Cancer Center

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with an endotracheal tube: Participants undergoing general anesthesia with an endotracheal tube will have a gastric tube blindly inserted by an anesthesia provider.
  Interventions: Other: Blind Gastric Tube Placement

INTERVENTIONS:
Other: Blind Gastric Tube Placement — The provider will be blinded to the ultrasound imaging throughout the entire insertion. This blind insertion process is the standard of care currently practiced at MSKCC. After the provider verbalizes that they have completed the insertion the investigators will stop the ultrasound imaging and complete the data form. No information will be given to the provider about the location of the gastric tube as to not deviate from the standard of care. The only time that information will be provided to the practitioner inserting the tube will be if the tube is positioned in any of the following positions that are thought to be potentially injurious if unrecognized. These positions include intrapulmonary, cranial, nasal or oral pharyngeal placements and diverticular or hiatal hernia sac coiling and remain unrecognized by the practitioner. These are considered positions that have the potential for injury and therefore will be divulged to prevent ensuing injury.

SUMMARY:
This is a prospective, single-arm cohort, observational study to determine the incidence of gastric tube malposition during blind insertion by an anesthesia provider.

ELIGIBILITY:
Inclusion Criteria:

* The adult population, ages 18 and greater
* Patients undergoing general anesthesia with an endotracheal tube that will have a gastric tube blindly inserted by an anesthesia provider

Exclusion Criteria:

* Pediatric population (<18 years)
* Gastric tube inserted under direct visualizing (the use of a Mac or Miller laryngoscope or any video laryngoscope)
* Inability to visualize gastric tube by ultrasound due to body habitus, analogous anatomy, etc
* Pre-anesthesia insitu gastric tube
* Gastric tube inserted by practitioner other than a member of the anesthesia team

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants undergoing general anesthesia with an endotracheal tube that will have a gastric tube blindly inserted by an anesthesia provider.
Sampling Method: Non-Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Incidence of malposition of blindly placed gastric tubes by anesthesia providers | Day of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Luis E Tollinche, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://mskcc.org